CLINICAL TRIAL: NCT06125860
Title: Targeting Strategies of Antenatal Balanced Energy and Protein Supplementation in Addis Ababa, Ethiopia
Brief Title: BEP Targeting Strategies in Ethiopia
Acronym: BEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Addis Continental Institute of Public Health (Other); George Mason University (Other)
Responsible Party: Principal Investigator, Wafaie Fawzi, Richard Saltonstall Professor of Population Sciences, and Professor of Nutrition, Epidemiology, and Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB22-1245
Record Dates: First submitted 2023-10-31; First posted 2023-11-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-01

CONDITIONS: Small for Gestational Age at Delivery; Gestational Weight Gain; Stillbirth; Preterm Birth; Birth Weight; Maternal Anemia in Pregnancy, Before Birth; Neonatal Death; Perinatal Death
Keywords: balanced energy and protein supplementation; food supplementation; antenatal nutrition; maternal nutrition; gestational weight gain; Ethiopia
MeSH Terms: conditions — Gestational Weight Gain; Stillbirth; Premature Birth; Birth Weight; Perinatal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (control arm) (No Intervention): In Arm 1 (control arm), participants will receive the standard of antenatal care including iron and folic acid supplementation.
- Arm 2 (Targeted BEP based on baseline nutritional status) (Experimental)
  Interventions: Dietary Supplement: Targeted BEP based on baseline nutritional status
- Arm 3 (Targeted BEP by baseline nutritional status and monthly gestational weight gain monitoring) (Experimental)
  Interventions: Dietary Supplement: Targeted BEP based on baseline nutritional status and monthly GWG monitoring
- Arm 4 (universal BEP) (Experimental)
  Interventions: Dietary Supplement: Universal BEP

INTERVENTIONS:
Dietary Supplement: Targeted BEP based on baseline nutritional status — In Arm 2 (targeted BEP based on baseline nutritional status), in addition to the standard of care, participants will receive BEP supplements if their baseline BMI is less than 18.5 or their baseline mid-upper arm circumference is less than 23 cm.
  Arms: Arm 2 (Targeted BEP based on baseline nutritional status)
Dietary Supplement: Targeted BEP based on baseline nutritional status and monthly GWG monitoring — In Arm 3 (targeted BEP based on baseline nutritional status and monthly GWG monitoring), in addition to the standard of care, participants will receive BEP supplements if their baseline BMI is less than 18.5 or their baseline mid-upper arm circumference is less than 23 cm; participants with an inadequate GWG at a monthly follow-up visit will receive additional BEP supplements.
  Arms: Arm 3 (Targeted BEP by baseline nutritional status and monthly gestational weight gain monitoring)
Dietary Supplement: Universal BEP — In Arm 4 (universal BEP), all participants will receive BEP supplements from baseline through the end of pregnancy.
  Arms: Arm 4 (universal BEP)

SUMMARY:
The goal of this randomized effectiveness study is to evaluate the different targeting strategies for the delivery of balanced energy and protein (BEP) supplements among pregnant women in Addis Ababa, Ethiopia. The main goals of the study are to: 1) determine the effectiveness of two individual-based antenatal BEP targeting strategies for preventing adverse pregnancy outcomes; 2) compare the cost-effectiveness of the universal BEP provision with two individual-based targeting strategies for preventing adverse pregnancy outcomes; and 3) generate implementation evidence regarding the feasibility and acceptability of different antenatal BEP targeting strategies. Pregnant women will be enrolled during pregnancy, assigned to different strategies of BEP supplementation, and followed from pregnancy through six weeks postpartum to evaluate the impacts of different BEP targeting strategies on pregnancy, maternal, and child outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant women aged 18 to 49;
2. attending antenatal visits in one of the study health facilities;
3. with a gestational age of 24 weeks or less;
4. no known allergies to peanuts or soybeans;
5. having resided in the current location for at least 6 months;
6. intending to continue antenatal follow-up in the health facility;
7. intending to give birth and remain in the study area until six weeks after delivery; and
8. willing to take the BEP supplements for the entire duration of the pregnancy if eligible.

Exclusion Criteria:

* Not meeting all of the inclusion criteria above

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6750 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Small-for-gestational-age births | Assessed within 72 hours of birth
  Live birth whose birthweight for sex and gestational age is < 10th percentile based on the INTERGROWTH-21st standards

SECONDARY OUTCOMES:
Inadequate gestational weight gain | At the last weight measurement before delivery, at around 36 weeks
  Gestational weight gain percent adequacy ratio less than 90% at the last weight measurement before delivery, based on the Institute of Medicine recommendations
Excessive gestational weight gain | At the last weight measurement before delivery, at around 36 weeks
  Gestational weight gain percent adequacy ratio greater than 125% at the last weight measurement before delivery, based on the Institute of Medicine recommendations
Stillbirth | Between 28 weeks of gestation and delivery
  Fetal death between 28 weeks of gestation and delivery
Preterm birth | Less than 37 completed weeks of gestation
  Live birth < 37 completed weeks of gestation
Low birthweight | Assessed within 72 hours of birth
  Live birth weighing < 2500 grams
Macrosomia | Assessed within 72 hours of birth
  Live birth weighing > 4000 grams
Large-for-gestational-age births | Assessed within 72 hours of birth
  Live birth whose birthweight for sex and gestational age is > 90th percentile based on the INTERGROWTH-21st standards
Third-trimester anemia | At 32 weeks of gestation
  Hemoglobin concentration < 11 g/dL at 32 weeks of gestation
Neonatal death | From birth through 28 days of life
  Death of live newborn < 28 days of life
Perinatal death | Between 28 weeks of gestation to 7 days after delivery
  Fetal death between 28 weeks gestational age and delivery, or newborn death < 7 days of life
Pre-eclampsia | After 20 weeks of gestation
  New onset hypertension (systolic blood pressure >= 140 or diastolic blood pressure >=90 mmhg) after 20 weeks of gestation with proteinuria.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, DrPH, MBBS, Principal Investigator — Harvard School of Public Health (HSPH); Yemane Berhane, MD, PhD, Principal Investigator — Addis Continental Institute of Public Health
Locations (1):
- Addis Continental Institute of Public Health (ACIPH), Addis Ababa, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang D, Shifraw T, Costa JC, Abdelmenan S, Tsegaye S, Berhane Y, Gulema H, Berhane H, Fasil N, Workneh F, Tarekegn W, Wang M, Menzies NA, Worku A, Berhane Y, Fawzi WW. Targeting strategies of antenatal balanced energy and protein supplementation in Addis Ababa, Ethiopia: study protocol for a randomized effectiveness study. Trials. 2024 Apr 30;25(1):291. doi: 10.1186/s13063-024-08002-2. PMID 38689304